CLINICAL TRIAL: NCT03711695
Title: Validation of Signal Waveforms in a Consumer-based Wristwatch Prototype Device During Standard Cardiac Procedures
Brief Title: iBeat Wristwatch Validation Study
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: iBeat Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 17-23761
Record Dates: First submitted 2018-02-27; First posted 2018-10-18 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Arrythmia, Cardiac
Keywords: ibeat; wrist watch; digital health; Arrythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (3):
- Group A: Subjects presenting for catheter ablation for cardiac arrhythmias (e.g. atrial fibrillation, supraventricular tachycardia, or ventricular tachycardia)
  Interventions: Device: iBeat wristwatch device
- Group B: Subjects judged based on the clinical evaluation of high, greater than 75%, atrial pacing or ventricular pacing burden or known pacing dependence with planned device interrogation for: 1) pacemaker (single or dual chamber), 2) implantable cardioverter-defibrillator (single or dual chamber), or 3) cardiac resynchronization therapy with or without defibrillator (single or dual chamber plus left ventricular pacing).
  Interventions: Device: iBeat wristwatch device
- Group C: Subjects for clinically indicated defibrillation threshold testing (DFT) (with a transvenous or subcutaneous implantable cardioverter defibrillator (ICD) lead system)
  Interventions: Device: iBeat wristwatch device

INTERVENTIONS:
Device: iBeat wristwatch device — The participant will be asked to wear one iBeat wristwatch device on each arm during the planned procedure.

SUMMARY:
The iBeat Study is a single-center, prospective, unblinded validation of the photoplethysmography (PPG) and tissue oximetry (TO) signal waveforms recorded from a wrist-based sensor devices.

DETAILED DESCRIPTION:
The goal of the proposed research is to validate PPG and TO signal waveforms recorded from a wist-based sensor device, which is worn on one or both arms, during catheter ablation, device interrogation, and defibrillation threshold testing (DFT). It is a non-invasive procedure that will include placing a wrist-based sensor on subjects who consent participate. Data collected from routine clinical care devices used during these procedures (catheter ablations, device interrogations, and DFTs) will confirm data collected from the iBeat wristwatch.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 years and ≤ 85 years
2. Able to understand and give informed consent.
3. Subject is presenting for the following planned procedures:

3.1 Group A (25 subjects): Subjects presenting for catheter ablation for cardiac arrhythmias (e.g. atrial fibrillation, supraventricular tachycardia, or ventricular tachycardia) 3.2 Group B (25 subjects): Subjects judged based on the clinical evaluation of high, greater than 75%, atrial pacing or ventricular pacing burden or known pacing dependence with planned device interrogation for: 1) pacemaker (single or dual chamber), 2) implantable cardioverter-defibrillator (single or dual chamber), or 3) cardiac resynchronization therapy with or without defibrillator (single or dual chamber plus left ventricular pacing).

3.3 Group C (5 subjects): Subjects for clinically indicated defibrillation threshold testing (DFT) (with a transvenous or subcutaneous ICD lead system)

Exclusion Criteria:

1. Age < 21 years and > 85 years
2. Unable to or refuse to give written informed consent
3. Unwilling or unable to wear the smartwatch device on at least one wrist
4. Uncorrected severe aortic stenosis or subaortic stenosis (including hypertrophic cardiomyopathy) with outflow tract obstruction > 50 mm
5. New York Heart Association Class IV Heart Failure

Ages: 21 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adults that present for either catheter ablation, cardiac device interrogation, or defibrillation threshold testing.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Detect hemodynamic significant (e.g. Ventricular tachycardia, ventircular fibrillatio, supra ventricular tachycardia with fast ventricular rate, etc) arrhythmias using photoplethysmography | Immediate
  Detect hemodynamic significant arrhythmia using changes in photoplethysmography [PPG] as measured using a wrist-watch.
Detect hemodynamic significant (e.g. Ventricular tachycardia, ventircular fibrillatio, supra ventricular tachycardia with fast ventricular rate, etc) arrhythmias using tissue oxygenation | Immediate
  Detect hemodynamic significant arrhythmia using changes in tissue oxygenation as measured using a wrist-watch.

SECONDARY OUTCOMES:
Detect benign arrhythmia (e.g. sinus tachycardia, atrial flutter, atrial fibrillation supra-ventricular tachycardia) using changes in photoplethysmography | Immediate
  Detect hemodynamic significant arrhythmia by using changes in photoplethysmography signal, as measured using a wrist-watch.
Detect benign arrhythmia (e.g. sinus tachycardia, atrial flutter, atrial fibrillation supra-ventricular tachycardia) using changes in tissue oxygenation | Immediate
  Detect hemodynamic significant arrhythmia by using changes in tissue oxygenation signal, as measured using a wrist-watch.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Olgin, MD, Principal Investigator — University of California, San Francisco; Robert Avram, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
The patient data will not be shared with other researchers. However, study outcomes will be published in peer-reviewed journals.